CLINICAL TRIAL: NCT03327454
Title: Non-Interventional Observational Study on Patient Satisfaction With the Benepali® Pre-Filled Pen
Brief Title: Benepali® PEN Patient Satisfaction Survey
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: GER-BNP-16-11103
Record Dates: First submitted 2017-10-11; First posted 2017-10-31 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Rheumatoid Arthritis; Spondyloarthropathies
Keywords: Ankylosing spondylitis; Axial spondyloarthritis; Benepali pen; Etanercept; Patient questionnaire; Pre-filled pen; Biological DMARDs; Antirheumatic drug
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthropathies; Spondylitis, Ankylosing; Axial Spondyloarthritis | interventions — Etanercept

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Benepali: Treatment of participants with the Benepali pre-filled pen takes place in accordance with the prescribing information and standard medical practice.
  Interventions: Biological: Benepali

INTERVENTIONS:
Biological: Benepali — Administered as specified in the treatment arm.
  Other Names: Etanercept

SUMMARY:
The main aim of this study is to ascertain general satisfaction among participants with rheumatic diseases with day-to-day use of the Benepali® prefilled pen by means of a standardised participant questionnaire. In addition, it is to be investigated whether differences exist in general participant satisfaction between participant groups who have undergone various prior treatment and/or have previous experience with application systems (participants new to the use of biologics, participants changing over from a prefilled injection or changing over from another pre-filled pen) and between participants of the various indication groups. Furthermore, the participants are to evaluate various aspects of using the Benepali® pre-filled pen based on their personal experience, such as e.g. handling, user-friendliness and features of the Benepali® pre-filled pen, as well as the effectiveness of the training on injection with the Benepali® pre-filled pen, based on participant satisfaction with the training received with the training pen and the evaluation of the training material received.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of moderate to severe active rheumatoid arthritis, severe active and progressive rheumatoid arthritis, active and progressive psoriatic arthritis, severe active ankylosing spondylitis, or severe non-radiographic axial spondyloarthritis
* Current treatment with the Benepali® pre-filled pen in accordance with prescribing information for at least 3 months beforehand
* The patient has signed a declaration of consent to take part in the study

Key Exclusion Criteria:

* Patients who are receiving Benepali® for the treatment of moderate to severe plaque psoriasis
* Patients who exhibit contraindications in accordance with the prescribing information for Benepali® and therefore treatment with Benepali ® is not indicated

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who are treated by practitioners in Germany and who are eligible according to the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2018-06-21 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants that are "Very Satisfied (4)" or "Satisfied (3)" with the Benepali Pre-Filled Pen | Day 1
  The Questionnaire is based on a 5-point Likert scale where 0 = very dissatisfied, 1 = dissatisfied, 2 = neither dissatisfied nor satisfied, 3 = satisfied, 4 = very satisfied.

SECONDARY OUTCOMES:
Percentage of Participants that Answered Questions on Their Personal Experience of Various Aspects of Using the Benepali Pre-Filled Pen with a (3) or (4) on a 5-point Likert Scale. | Day 1
  The questions comprise the areas of handling, user-friendliness and features of the Benepali® pre-filled pen, satisfaction compared with the previous application system and satisfaction with the training on injection with the training pen. 0 = worst rating, 4 = best rating.
Percentage of Participants that Answered "Yes" in Terms of Satisfaction with Training Materials | Day 1
  The participants evaluated the training materials and answered "yes" or "no" to questions regarding the adequate effectiveness, clarity, and extent of information provided.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (32):
- Germany (32):
  - Research Site, Altenholz
  - Research Site, Bad Neuenahr-Ahrweiler
  - Research Site, Berlin
  - Research Site, Braunschweig
  - Research Site, Coburg
  - Research Site, Cologne
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Ehringshausen
  - Research Site, Erfurt
  - Research Site, Essen
  - Research Site, Giessen
  - Research Site, Göpping
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Homburg
  - Research Site, Jülich
  - Research Site, Kronach
  - Research Site, Leipzig
  - Research Site, Ludwigshafen
  - Research Site, Magdeburg
  - Research Site, Mansfeld
  - Research Site, Mittelherwigsdorf
  - Research Site, München
  - Research Site, Neuss
  - Research Site, Norderstedt
  - Research Site, Nuremberg
  - Research Site, Offenberg
  - Research Site, Saarbrücken
  - Research Site, Seesen
  - Research Site, Tübingen
  - Research Site, Ulm

IPD SHARING:
Plan to Share IPD: No